CLINICAL TRIAL: NCT02135913
Title: Roles of Vitamin D and HDL in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang-An Li (Other)
Responsible Party: Sponsor-Investigator, Xiang-An Li, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-0348-P3H
Record Dates: First submitted 2014-04-25; First posted 2014-05-12 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Obese; Vitamin D Deficiency; Low HDL
Keywords: Obese; Children; Vitamin D deficiency; Low HDL
MeSH Terms: conditions — Obesity; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Viatamin D (Experimental): All children enrolled into the study will be prescribed standard of care vitamin D.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — All subjects enrolled into the study will be prescribed standard of care Vitamin D

SUMMARY:
This is a pilot study to determine the association between Vitamin D deficiency in obese children and low high density lipoprotein (HDL) and dysfunctional HDL.

DETAILED DESCRIPTION:
Subjects will be identified through the Department of Pediatric - High Body Mass Index (BMI) Clinic by Dr. Aurelia Radulescu during standard of care visit. Dr. Radulescu will determine if the subject meets study eligibility requirements.

Visit 1 (Baseline/Screening): Consent/assent will be obtained, medical history, demographic information along with height and weight will be collection. Clinical Laboratory testing, although not part of this study, will include the following standard of care tests. The results of Vitamin D and Lipid profile testing will be shared with Dr. Li by Dr. Radulescu.

* Lipid profile
* Vitamin D
* AST/ALT
* Hb A1C
* Glucose
* CBS w/diff
* TSH
* BUN, Creatine
* UA

Subjects will be placed on standard of care Vitamin D supplementation for 12 weeks.

Visit 2 (3 month visit) End of Study: Subjects will return to the BMI clinic at month 3 for follow-up and additional clinical laboratory testing (see visit 1 for a description of testing to be performed) in order to assess their response to Vitamin D supplementation. Subjects with previously reported abnormal Lipid values will have a Lipid profile repeated at this visit. Month 3 visit will be the End of Study visit.

ELIGIBILITY:
Inclusion Criteria:

* Obese children
* Vitamin D deficiency
* Low HDL

Exclusion Criteria:

* HIV
* Hepatitis A
* Hepatitis B
* Hepatitis C
* Non-English speaking

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Laboratory Analysis of Vitamin D blood levels before Vitamin D Supplementation | up to 24 months
  Vitamin D deficiency in obese child leads to low HDL and dysfunctional HDL

SECONDARY OUTCOMES:
Laboratory Analysis of Vitamin D Blood Levels following Vitamin D Supplementation | up to 24 months
  Supplementation of Vitamin D to obese children with low Vitamin D/low HDL corrects Vitamin D deficiency, restores HDL levels and functions.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang An-Li, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States